CLINICAL TRIAL: NCT06719362
Title: A First-in-human, Open-label, Dose Escalation, Phase I Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Clinical Efficacy of M3T01 Monotherapy and in Combination With Pembrolizumab and Other Systemic Therapies in Patients With Advanced Solid Tumors
Brief Title: A Clinical Trial to Evaluate the Safety, Tolerability and Clinical Efficacy of M3T01 Monotherapy and in Combination With Pembrolizumab and Other Systemic Therapies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024000813
Record Dates: First submitted 2024-11-21; First posted 2024-12-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab; Chemoradiotherapy; Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1A: DL 1 (Experimental): M3T01 100 mg as monotherapy.
  Interventions: Drug: M3T01
- Part 1A: DL 2 (Experimental): M3T01 200 mg as monotherapy.
  Interventions: Drug: M3T01
- Part 1A: DL 3 (Experimental): M3T01 400 mg as monotherapy.
  Interventions: Drug: M3T01
- Part 1A: DL 4 (Experimental): M3T01 600 mg as monotherapy.
  Interventions: Drug: M3T01
- Part 1A: DL 5 (Experimental): M3T01 800 mg as monotherapy.
  Interventions: Drug: M3T01
- Part 1B: DL 6 (Experimental): M3T01 400 mg in combination with pembrolizumab 200 mg.
  Interventions: Drug: M3T01; Drug: Pembrolizumab
- Part 1B: DL 7 (Experimental): M3T01 600 mg in combination with pembrolizumab 200 mg.
  Interventions: Drug: M3T01; Drug: Pembrolizumab
- Part 1B: DL 8 (Experimental): M3T01 800 mg in combination with pembrolizumab 200 mg.
  Interventions: Drug: M3T01; Drug: Pembrolizumab
- Part 2A: Newly diagnosed glioblastoma with unmethylated MGMT promoter (Experimental): Subjects will be treated with standard of care chemoradiation therapy consisting of TMZ 75 mg/m2 daily with concurrent radiation therapy (60 Gy administered over 6 weeks). Following chemoradiation therapy, subjects will have a 4-week break from TMZ before starting standard adjuvant TMZ 150-200 mg/m2 days 1-5 of 28-day cycles for 6 cycles. Subjects will be treated with M3T01 at the RP2D through an IV infusion every 3 weeks that will begin concurrently with chemoradiation therapy.
  Interventions: Drug: M3T01; Radiation: Chemoradiation
- Part 2B: First-line tx for unresectable/metastatic HER2- esophageal, GEJ, or gastric adenocarcinoma. (Experimental): Subjects with unresectable or metastatic HER2 negative esophageal, gastroesophageal (GEJ), or gastric adenocarcinoma without prior systemic therapy in the metastatic setting will be treated with M3T01 at the RPD2 in combination with standard of care pembrolizumab plus FOLFOX chemotherapy.
  Interventions: Drug: M3T01; Drug: Pembrolizumab; Drug: FOLFOX regimen
- Part 2C: Second-line treatment for recurrent/metastatic HNSCC (Experimental): Subjects with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) who have developed disease progression after first-line systemic therapy with an anti-PD-1-based regimen in the recurrent or metastatic setting will be treated with M3T01 at the RP2D in combination with pembrolizumab 200 mg IV every 3 weeks for up to 2 years.
  Interventions: Drug: M3T01; Drug: Pembrolizumab

INTERVENTIONS:
Drug: M3T01 — Subjects will be treated with M3T01 through an IV infusion over 1 hour given every 3 weeks.
Drug: Pembrolizumab — Pembrolizumab will be given as standard of care to Cohort DL 5+ under Part 1 of the study. Subjects will receive 200 mg IV once every 3 weeks.
  Other Names: KEYTRUDA
  Arms: Part 1B: DL 6; Part 1B: DL 7; Part 1B: DL 8; Part 2B: First-line tx for unresectable/metastatic HER2- esophageal, GEJ, or gastric adenocarcinoma.; Part 2C: Second-line treatment for recurrent/metastatic HNSCC
Radiation: Chemoradiation — Subjects will be treated with standard of care chemoradiation therapy consisting of TMZ 75 mg/m2 daily with concurrent radiation therapy (60 Gy administered over 6 weeks). Following chemoradiation therapy, subjects will have a 4-week break from TMZ before starting standard adjuvant TMZ 150-200 mg/m2 days 1-5 of 28-day cycles for 6 cycles. Subjects will be treated with M3T01 at the RP2D through an IV infusion every 3 weeks that will begin concurrently with chemoradiation therapy.
  Arms: Part 2A: Newly diagnosed glioblastoma with unmethylated MGMT promoter
Drug: FOLFOX regimen — FOLFOX will be given as standard of care on 14 day cycles. Subjects will receive oxaliplatin 85 mg/m2 IV on Day 1, leucovorin 400 mg/m2 IV on Day 1, fluorouracil 400 mg/m2 IV push on Day 1, and fluorouracil 1,200 mg/m2 IV continuous infusion on Days 1-2 every 14 days for up to 9 cycles.
  Other Names: Oxaliplatin, Leucovorin, Fluorouracil
  Arms: Part 2B: First-line tx for unresectable/metastatic HER2- esophageal, GEJ, or gastric adenocarcinoma.

SUMMARY:
Phase 1 first-in-human, open-label, dose-escalation (3 + 3), dose-expansion clinical trial to evaluate the safety, tolerability and preliminary clinical efficacy of M3T01 (fully human IgG4/kappa monoclonal antibody targeting FasL) in subjects with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, phase I, open-label, dose escalation, dose expansion clinical trial designed to evaluate the safety, tolerability and preliminary clinical efficacy of M3T01 monotherapy and in combination with standard of care systemic therapies (including pembrolizumab, temozolomide, and FOLFOX) in subjects with advanced solid tumors. Within the Part 1 dose escalation stage of the study, the maximum tolerated dose (MTD) or maximum administered dose (MAD) for M3T01 monotherapy and in combination with pembrolizumab will be determined. The recommended phase 2 dose (RP2D) will be determined based upon available pharmacokinetic, pharmacodynamic, and preliminary clinical efficacy data and will be equal to or lower than the MTD. M3T01 will be administered at the RP2D in combination with standard of care systemic therapies (including pembrolizumab, temozolomide, and FOLFOX) in the Part 2 dose expansion stage of the clinical trial.

Up to 48 subjects will be enrolled in the Part 1 dose escalation stage of the study (depending on observed toxicity and when the MTD/MAD is reached). The Part 2 dose expansion portion of the study will enroll up to 62 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Life expectancy ≥ 12 weeks.
3. Provision of written informed consent (see Section 16.1 and Appendix 18.5.5) for participation in the clinical trial.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1 for subjects with solid tumors other than glioblastoma.
5. Karnofsky Performance Status of ≥ 70% for subjects with glioblastoma.
6. Tumor tissue from a surgical or core needle biopsy must be provided to the sponsor (fine needle aspirate or cytology specimens are not acceptable). Archival formalin fixed paraffin embedded (FFPE) tissue is acceptable. If archival tumor tissue is not available, a fresh tumor biopsy must be performed.
7. Subjects must have a tumor accessible for biopsy while on treatment. If the subject does not have a tumor that is safely accessible for biopsy, the subject may still participate in the clinical trial following authorization from the sponsor. NOTE: Subjects with glioblastoma are not required to have tumor accessible for biopsy and will not undergo a protocol specified biopsy on study.
8. Eligible tumor types in Part 1 Dose Escalation will include subjects with histologically or cytologically confirmed metastatic or unresectable solid tumors who have developed disease progression following standard systemic therapy in the unresectable or metastatic setting. Subjects with cancers that harbor a molecularly defined oncogenic target for which an FDA approved therapy is available (including but not limited to EGFR, ROS1, ALK, BRAF, RET, NTRK, KRAS G12C, etc.) should have received this therapy.
9. Measurable disease

   * Subjects with solid tumors other than glioblastoma must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
   * Subjects with glioblastoma: Part 1: must have measurable disease per Response Assessment in Neuro-Oncology (RANO 2.0); Part 2: measurable disease at baseline is not required as these subjects will have undergone maximal safe resection prior to enrollment.
10. Adequate organ function as defined by the following:

    * Absolute neutrophil count (ANC) ≥ 1.2 x 109/L.
    * Hemoglobin ≥ 9.0 g/dL (without a blood transfusion 2 weeks prior to the hemoglobin measurement).
    * Platelet count ≥ 100 x 109/L (without a platelet transfusion 2 weeks prior to the platelet measurement).
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN.
    * Total bilirubin ≤ 1.5 x ULN (or ≤ 3 x ULN for subjects with Gilbert's syndrome).
    * International normalized ratio (INR) ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (unless the subject is being treated with anticoagulant medication).
    * Serum albumin ≥ 2.8 g/dL.
    * Creatinine clearance (measured or calculated) ≥ 30 mL/min.
11. Female subjects of reproductive potential who are sexually active with a male partner must:

    * Have a negative serum beta-human chorionic gonadotropin (β-HCG) test within 3 days of cycle 1 day 1.
    * Agree to use highly effective contraceptive measures (as defined in protocol) from the time of enrollment through 3 months after the last dose of study drug in the clinical trial.
    * Female subjects are considered to be of non-reproductive potential if they: have been amenorrheic for greater than 1 year or have undergone surgical sterilization through tubal ligation, oophorectomy or hysterectomy.
12. Male subjects with a female partner of reproductive potential must agree to use highly effective contraception (as defined in protocol) from the time of enrollment through 3 months after the last dose of study drug administration.
13. Subjects must agree to not donate sperm or eggs (ova, oocytes) for the purpose of reproduction from the time of enrollment through 3 months after the last dose of study drug administration.
14. Toxicities from prior anti-cancer therapy must have resolved to grade ≤ 1.

    * Exceptions include vitiligo, endocrinopathies managed with hormone replacement therapy, alopecia, and grade 2 neuropathy or hearing loss.

Exclusion Criteria:

1. Treatment with anticancer therapy within 14 days or 5 half-lives (whichever is shorter) of cycle 1 day 1. Palliative radiation therapy to a non-CNS metastasis is permitted if completed at least 14 days prior to cycle 1 day 1.
2. History of other active malignancy that required treatment within 2 years of enrollment. Exceptions include the following:

   * Early-stage/localized tumors that have received definitive/curative treatment and have low risk of recurrence (including but not limited to cutaneous squamous cell or basal cell carcinoma, in situ cervical or bladder cancer, and early-stage prostate cancer).
   * Early-stage prostate cancer in which observation without treatment is recommended.
3. Clinically significant cardiovascular conditions as defined by the following:

   * New York Heart Association (NYHA) congestive heart failure class ≥ II.
   * Left ventricular ejection fraction ≤ 50%.
   * Clinically significant cardiac arrhythmia requiring treatment within 3 months of enrollment. Subjects with cardiac arrhythmias on stable management for over 3 months prior to enrollment are permitted.
   * Prolonged QTcF interval > 480 ms.
   * Myocardial infarction, stroke, or pulmonary embolism within 3 months of enrollment.
4. CNS metastases or leptomeningeal carcinomatosis (applicable to subjects with solid tumors other than glioblastoma). Subjects with brain metastases are eligible for participation if one of the following criteria are met:

   * CNS metastases have been treated with surgical resection or radiation therapy and have remained stable for at least 4 weeks (repeat imaging required at least 4 weeks following resection or last radiation therapy) prior to cycle 1 day 1.
   * The subject is neurologically asymptomatic and there are ≤ 4 CNS metastases no larger than 1 cm.
5. Treatment with immunosuppressive medications.

   - Treatment with corticosteroids greater than the equivalent of prednisone 10 mg/day within 2 weeks of cycle 1 day 1 is exclusionary. Exceptions include: Premedication with corticosteroids for iodine contrasted CT scans; Chronic use of ≤ 10 mg/day of prednisone (or equivalent). Topical, inhaled, and intra-articular corticosteroid use is allowed; Subjects with glioblastoma are permitted to be on ≤ 3 mg/day dexamethasone (or equivalent).
6. History of severe pulmonary disease defined as either of the following:

   * History of interstitial lung disease, non-infectious pneumonitis (including immune checkpoint inhibitor induced pneumonitis), or pulmonary fibrosis.
   * Currently dependent on supplemental oxygen.
7. History of allogeneic stem cell or solid organ transplantation.
8. History of autoimmune disease that required systemic immunosuppressive therapy within 2 years of enrollment. Subjects with autoimmune diseases managed with hormone replacement or topical therapies are eligible.
9. History of an immune-mediated adverse event from treatment with an immune checkpoint inhibitor that resulted in treatment discontinuation.

   - Subjects who discontinued treatment with ipilimumab due to toxicity and subsequently tolerated treatment with an anti-PD-(L)1 inhibitor without treatment-limiting toxicity are eligible.
10. History of severe hypersensitivity reaction (≥ grade 3) to infusion of a therapeutic monoclonal antibody.
11. Any major surgery within 4 weeks of receiving the first dose of the investigational treatment.
12. Women who are pregnant or breast feeding.
13. Subjects with active (acute or chronic) bacterial, viral, or fungal infection at the time of enrollment are ineligible with the following exceptions:

    * Subjects with human immunodeficiency virus (HIV) are eligible for participation if the following criteria are met: CD4+ T cell count ≥350 cells/µL, No history of AIDS-defining opportunistic infections within 12 months of enrollment, Subjects must be on antiretroviral therapy for at least 4 weeks and have an HIV viral load less than 400 copies/mL prior to enrollment.
    * Subjects with chronic hepatitis B (HBV) who are on suppressive antiviral therapy prior to enrollment are eligible. Subjects with chronic HBV who are not eligible for treatment with suppressive antiviral therapy are ineligible.
    * Subjects with a history of hepatitis C (HCV) infection who have completed curative antiviral treatment and have an HCV viral load below the limit of quantification are eligible.
14. Ongoing drug or alcohol abuse at the time of enrollment.
15. Any medical or psychiatric illness or social circumstance that could jeopardize compliance with the protocol directed treatment and safety assessments.

Additional Exclusion Criteria Specific for the Part 2A - Newly Diagnosed MGMT Unmethylated Glioblastoma Cohort:

1. Subjects with recurrent or secondary GBM.
2. Subjects who underwent biopsy only without maximal safe resection.
3. Subjects with a contraindication to MRI scans.
4. Subjects with IDH-1 or IDH-2 mutations or H3 K27M diffuse midline glioma.
5. Subjects with unresolved CNS hemorrhage, leptomeningeal or spinal metastases or ventricular invasion.
6. Subjects treated with a carmustine wafer implant.
7. Subjects treated with Tumor Treating Fields (TTF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 4 years
  Safety parameters including clinical assessments, vital signs, laboratory testing, and electrocardiograms (ECG) will be used to assess treatment-emergent adverse events (TEAE). Adverse events will be graded using the NCI-CTCAE v5.0. Investigators will determine relatedness of all treatment emergent adverse events (TEAE) to the investigational agent(s).
Dose-limiting toxicities | 21 days after C1D1
  The DLT evaluation period will be defined as the first 21 days after infusion of M3T01 as monotherapy or in combination with other systemic therapies (including pembrolizumab, temozolomide, and FOLFOX). Site investigators will grade toxicities using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Serious adverse events | 4 years
  Clinical assessments, vital signs, laboratory testing, and electrocardiograms (ECG) will be used to assess serious adverse events (SAE) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Immune-related adverse events | 4 years
  Clinical assessments, vital signs, laboratory testing, and electrocardiograms (ECG) will be used to assess immune-related adverse events (irAE) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
PK Profile of M3T01 | 4 years
  Serum PK parameters including the area under the curve (AUC), maximum concentration (Cmax), minimum concentration (Cmin), time to maximum concentration (Tmax), half-life (t1/2), and other serum concentration vs time parameters.
Immunogenicity of M3T01 | 4 years
  • Incidence of anti-drug antibodies (ADA) and neutralizing antibodies (nAbs) against M3T01 and correlation with M3T01 PK parameters, toxicity, and clinical efficacy.
Antitumor Activity of M3T01 | 4 years
  Tumor response (for all solid tumors other than glioblastoma) will be evaluated by site investigators per RECIST v1.1 to assess the objective response rate (ORR), best overall response (BOR), disease control rate (DCR), duration of response (DOR), progression free survival (PFS), and overall survival (OS). Tumor assessment CT or MRI scans will be performed every 8 weeks for the first 6 months and then every 12 weeks thereafter. Tumor assessments for subjects with glioblastoma will be performed with contrast-enhanced MRI per the Response Assessment in Neuro-Oncology (RANO 2.0) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rom Leidner, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Cancer Institute - Franz Clinic, Portland, Oregon, United States